CLINICAL TRIAL: NCT04651400
Title: Multinational, Observational, Retrospective Study to Evaluate Coagulation Changes and the Influence of Antithrombin III Treatment in Patients With Severe COVID-19 Infection
Brief Title: Observational, Retrospective Study to Evaluate Coagulation Changes and the Influence of Antithrombin III Treatment in Patients With Severe COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: ATN105
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Antithrombin III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- COVID-19 patients who had received treatment with ATIII: Patient records of patients hospitalised for severe COVID-19 infection until 01.06.2020 that required oxygen therapy will be used to retrospectively gather baseline demographic data (age, gender, height, weight, ethnicity/race, blood group, rhesus factor) and comorbidities. Records will also be used to retrospectively gather information on routine coagulation and laboratory parameters measured as per local protocols (including where available: AT, aPTT, PT, Quick, INR, , fibrinogen, D-dimers, haemoglobin levels, and platelet count), and thromboembolic complications and bleeding events that occurred during the individual observational treatment period. Patients will be grouped into 2 cohorts; those that received treatment with ATIII and those that did not. ATIII was administered as per local guidelines at each institute.
  Interventions: Drug: Antithrombin III
- COVID-19 patients who had not received treatment with ATIII: Patient records of patients hospitalised for severe COVID-19 infection until 01.06.2020 that required oxygen therapy will be used to retrospectively gather baseline demographic data (age, gender, height, weight, ethnicity/race, blood group, rhesus factor) and comorbidities. Records will also be used to retrospectively gather information on routine coagulation and laboratory parameters measured as per local protocols (including where available: AT, aPTT, PT, Quick, INR, , fibrinogen, D-dimers, haemoglobin levels, and platelet count), and thromboembolic complications and bleeding events that occurred during the individual observational treatment period. Patients will be grouped into 2 cohorts; those that received treatment with ATIII and those that did not. ATIII was administered as per local guidelines at each institute.
- Non-COVID-19 patients who had received treatment with ATIII: A control group will be used to gather comparative data in non-COVID-19 patients.
  Data will be gathered retrospectively from patient records for severely ill patients who received oxygen therapy for non-COVID-19 infection until end 2019 (31.12.2019). Control group will also be grouped into 2 cohorts for those having received/ having not received ATIII treatment.
  Interventions: Drug: Antithrombin III
- Non-COVID-19 patients who had not received treatment with ATIII: A control group will be used to gather comparative data in non-COVID-19 patients.
  Data will be gathered retrospectively from patient records for severely ill patients who received oxygen therapy for non-COVID-19 infection until end 2019 (31.12.2019). Control group will also be grouped into 2 cohorts for those having received/ having not received ATIII treatment.

INTERVENTIONS:
Drug: Antithrombin III — Antithrombin III
  Groups: COVID-19 patients who had received treatment with ATIII; Non-COVID-19 patients who had received treatment with ATIII

SUMMARY:
Multicentre, multinational, non-interventional, observational, retrospective, patient record study to evaluate changes in coagulation parameters in patients with severe COVID-19 infection receiving/not treatment with antithrombin (AT) III

ELIGIBILITY:
For Sites in Austria:

Inclusion Criteria:

For the +COVID-19 group:

* Confirmed COVID-19 positive test result OR extremely high likelihood of COVID-19 infection (e.g., family member or other person co-habiting with subject with a documented infection; passenger from cruise ship with +COVID- 19)
* Hospitalisation for severe COVID-19 infection until 01.06.2020
* COVID-19 patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

For the control group:

* Hospitalisation for any disease other than COVID-19 infection until end 2019 (31.12.2019)
* Patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

Exclusion Criteria:

* Known hypersensitivity or allergic reaction to ATIII
* Participation in any interventional trial during the time of individual observational period (date of hospitalisation to the date of removal of oxygen therapy or death, whichever occurred first)
* Pregnant women

For Sites in France:

Inclusion Criteria:

For the +COVID-19 group:

* Confirmed COVID-19 positive test result OR extremely high likelihood of COVID-19 infection (e.g., family member or other person co-habiting with subject with a documented infection; passenger from cruise ship with +COVID-19)
* Hospitalisation for severe COVID-19 infection and discharged from the hospital or died before start of documentation. COVID-19 patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

For the control group:

* Hospitalisation for any disease other than COVID-19 infection until end 2019 (31.12.2019)
* Patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

Exclusion Criteria:

* Known hypersensitivity or allergic reaction to ATIII
* Participation in any interventional trial during the time of individual observational period (date of hospitalisation to the date of removal of oxygen therapy or death, whichever occurred first)
* Pregnant women

For sites in Germany:

Inclusion Criteria:

For the +COVID-19 group:

* Confirmed COVID-19 positive test result OR extremely high likelihood of COVID-19 infection (e.g., family member or other person co-habiting with subject with a documented infection; passenger from cruise ship with +COVID-19)
* Hospitalisation for severe COVID-19 infection until 01.02.2021.
* COVID-19 patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

For the control group:

* Hospitalisation for any disease other than COVID-19 infection until end 2019 (31.12.2019)
* Patients having required oxygen therapy as per local guidelines (including those requiring a ventilator, central venous catheter or ECMO)

Exclusion Criteria:

* Known hypersensitivity or allergic reaction to ATIII
* Participation in any interventional trial during the time of individual observational period (date of hospitalisation to the date of removal of oxygen therapy or death, whichever occurred first)
* Pregnant women

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A target of 150 patients (male and female) hospitalised with severe COVID-19 infection and having required oxygen therapy (including those requiring a ventilator, central venous catheter or ECMO) will be included into this study. A control group of matched numbers of non-COVID-19 patients hospitalised and having required oxygen therapy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Antithrombin Levels | throughout hospitalization, approximately 1-3 weeks
  Levels of AT in severely ill COVID-19 positive patients receiving/not receiving ATIII treatment

SECONDARY OUTCOMES:
aPPT Levels | throughout hospitalization, approximately 1-3 weeks
  aPPT Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
PT Levels | throughout hospitalization, approximately 1-3 weeks
  PT Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
Quick Levels | throughout hospitalization, approximately 1-3 weeks
  Quick Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
INR Levels | throughout hospitalization, approximately 1-3 weeks
  INR Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
D-dimer Levels | throughout hospitalization, approximately 1-3 weeks
  D-dimer Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
Fibrinogen Levels | throughout hospitalization, approximately 1-3 weeks
  Fibrinogen Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
Haemoglobin Levels | throughout hospitalization, approximately 1-3 weeks
  Haemoglobin Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
Platelet Levels | throughout hospitalization, approximately 1-3 weeks
  Platelet Levels in severely ill COVID-19 patients receiving/not receiving ATIII treatment and compared to control group
Thromboembolic complications and bleeding events between groups | throughout hospitalization, approximately 1-3 weeks
  Comparison of the occurrence of thromboembolic complications and bleeding events between groups
Comparison of the duration of requirement for oxygen therapy, and invasive ventilation support or ECMO between groups | throughout hospitalization, approximately 1-3 weeks
  Comparison of the duration of requirement for oxygen therapy, and invasive ventilation support or ECMO between groups
Hospital length of stay | throughout hospitalization, approximately 1-3 weeks
  Hospital length of stay between groups
Number of days in ICU | throughout hospitalization, approximately 1-3 weeks
  Number of days in ICU between groups
Number of days requiring oxygenation | throughout hospitalization, approximately 1-3 weeks
  Number of days requiring oxygenation between groups
Discharge disposition | throughout hospitalization, approximately 1-3 weeks
  Discharge disposition between groups
Mortality | throughout hospitalization, approximately 1-3 weeks
  Mortality between groups

CONTACTS AND LOCATIONS:
Locations (6):
- Austria (2):
  - Octapharma Research Site, Innsbruck
  - Octapharma Research Site, Vienna
- Octapharma Research Site, Strasbourg, France
- Germany (2):
  - Octapharma Research Site, Aachen
  - Octapharma Research Site, Essen
- ECMO Centre Karolinska, Stockholm, Sweden